CLINICAL TRIAL: NCT01788709
Title: PEG-Electrolyte Solution (FORTRANS®) With Mentholyptus Drops (Halls®) Versus Reduced Volume Ascorbic Acid Supplemented PEG-Electrolyte (MoviPrep®) in Colonoscopy Preparation: A Randomised Controlled Study
Brief Title: PEG-Electrolyte Solution (FORTRANS®) With Mentholyptus Drops (Halls®) Versus Reduced Volume Ascorbic Acid Supplemented PEG-Electrolyte (MoviPrep®) in Colonoscopy Preparation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: IM.AS1.32
Record Dates: First submitted 2013-02-08; First posted 2013-02-11 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2013-01

CONDITIONS: Bowel Cleansing in Preparation for Colonoscopy
Keywords: colonoscopy; preparation
MeSH Terms: interventions — MoviPrep

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Fortrans (split dose) + Mentholyptus drops
  Interventions: Other: preparation cleaning solution
- B (Active Comparator): MoviPrep (split dose)
  Interventions: Other: preparation cleaning solution

INTERVENTIONS:
Other: preparation cleaning solution
  Other Names: Fortrans (split dose) + Mentholyptus drops; MoviPrep (split dose)

SUMMARY:
The colonoscopy accuracy and safety depend on the quality of colon cleansing. An inadequately prepped bowel will increase the risk of missing a lesion, prolong procedure, increase patient discomfort, and eventually increase complication rate. Therefore an excellent colon cleansing is of extreme importance to the endoscopist and the patient.

Split Fortrans® prep with sugar-free mentholyptus drops (Halls®) has a better palatability and tolerability than the reduced volume ascorbic acid-supplemented PEG-electrolyte (MoviPrep®) in bowel cleansing for colonoscopy.

DETAILED DESCRIPTION:
Abstract:

Colorectal cancer is amongst the leading cancers worldwide. Treatment is greatly dependent on the stage of illness, with more favorable outcomes associated with early cancers. For this reason, screening colonoscopies have been increasing, as are efforts to improve the quality of bowel preparations. The colonoscopy accuracy and safety depend on the quality of colon cleansing. An inadequately prepped bowel will increase the risk of missing a lesion, prolong procedure, increase patient discomfort, and eventually increase complication rate. Hence, an Ideal bowel cleansing solution would quickly and reliably clean the colon while having a good tolerability and palatability to the patient. Current colonoscopy preparation regimens require the use of large volume of iso-osmotic PEG-electrolyte solution for adequate cleansing and are often poorly tolerated by patients. We have shown previously that mentholyptus drops significantly improved the palatability of PEG-electrolyte (Fortrans®) solution and the quality of preparation (1). We aim at this study to compare the efficacy of the above-mentioned prep technique and the reduced volume ascorbic acid-supplemented PEG-electrolyte (MoviPrep®). This is a randomized controlled trial that will include patients undergoing elective colonoscopy at the American University of Beirut Medical Center. Patients will be randomized into one of two study arms using a computer generated randomization list. 100 Patients will be asked to have candy (Halls®) during the whole 2 hours period while drinking the PEG solution (Fortrans®). Another 100 patients will be asked to take reduced volume ascorbic acid-supplemented PEG-electrolyte (MoviPrep®). All patients will then be interviewed by the research coordinator to evaluate the tolerability of the preparation while taking into account the palatability of the solution as main outcome and the remaining volume of the PEG solution and side effects as secondary outcomes. Based on the results of a pilot study, our sample size calculation showed that 100 patients per arm will be enough to attain significance. As for the statistical analysis, SPSS version 20.0 will be used for data entry and analysis.

I- Aim:

To compare the efficacy of split PEG-electrolyte (Fortrans®) with mentholyptus (Halls®) drops and the reduced volume ascorbic acid-supplemented PEG-electrolyte (MoviPrep®) in improving the palatability of solution used in bowel cleansing for colonoscopy.

II- Background:

The colonoscopy accuracy and safety depend on the quality of colon cleansing. An inadequately prepped bowel will increase the risk of missing a lesion, prolong procedure, increase patient discomfort, and eventually increase complication rate. Therefore an excellent colon cleansing is of extreme importance to the endoscopist and the patient. Hence, An Ideal bowel cleansing solution would quickly and reliably clean the colon while having a good tolerability and palatability to the patient. Poor tolerability by the patient would increase the risk of not finishing the whole solution and hence the risk of having a poor colon cleansing. Many types of bowel cleansing solutions are currently available in the market. Current colonoscopy preparation regimens require the use of large volume of iso-osmotic PEG-electrolyte solution for adequate cleansing and are often poorly tolerated by patients. Therefore, improving the tolerability of the solution by patients is of critical importance. The main side effects of bowel cleansing solution are nausea, vomiting, bloating, and cramps. To decrease their incidence and therefore to improve tolerability, one could either decrease the volume of the solution or improve its palatability. Many studies have tried to decrease the volume of the solution below the standard 4 liters. These studies have largely shown that smaller volume preps are inferior to standard preps. In addition, few studies have shown that improving palatability by adding a flavor improved patients' acceptance of the solution (2-6). MoviPrep® is the only liquid PEG bowel cleansing agent that incorporates ascorbic acid in its formulation, thus contributing to its lemon taste and consequently better patient tolerability. We have proved earlier this year through a randomized trial a high palatability of and hence a better quality of preparation (90% Good/Excellent) using the PEG-electrolyte Fortrans® with sugar-free mentholyptus drops (Halls®) (6).

We aim at comparing the colonoscopy preparation quality and the palatability of our technique and that of the MoviPrep® through a single blinded randomized trial.

III- Hypothesis:

Split Fortrans® prep with sugar-free mentholyptus drops (Halls®) has a better palatability and tolerability than the reduced volume ascorbic acid-supplemented PEG-electrolyte (MoviPrep®) in bowel cleansing for colonoscopy.

IV- Setting:

Single university based center (American University of Beirut Medical Center)

V- Study Design:

Prospective randomized single-blinded study

VI- Methods:

1. Study population:

   1. Inclusion criteria:

      ● Elective colonoscopy
      * Consent to the study
   2. Exclusion criteria:

      ● Pregnant or lactating women

      ● Age less than 18 years

      ● Significant gastroparesis

      ● Gastric outlet obstruction

      ● Ileus

      ● Known or suspected bowel obstruction or perforation

      ● Phenylketonuria
      * Glucose-6-phosphate dehydrogenase deficiency
      * Severe chronic renal failure (creatinine clearance <30 mL/minute)
      * Severe congestive heart failure (New York Heart Association [NYHA] class III or IV)
      * Dehydration
      * Severe acute inflammatory disease
      * Compromised swallowing reflex or mental status
      * Uncontrolled hypertension (systolic blood pressure ≥170 mm Hg, diastolic blood pressure ≥100 mm Hg)
      * Toxic colitis or megacolon

      These exclusion criteria are consistent with contraindications of currently approved bowel preparations; therefore, the results of this study may be generalized to the entire target population of patients undergoing colonoscopy, including the elderly.
2. Randomization:

   Patients will be enrolled by the principal investigator or study coordinator (MD) after assessing for inclusion and exclusion criteria. Patients will then be randomized into one of the two study arms using a pre-set randomization list where patients with an odd number as the last digit of their medical record will be assigned to the control arm and patients with an even number will be assigned to the intervention arm.
3. Study arms:

   ● First arm: 4 Liters of PEG solution (FORTRANS®) split into 2 days with sugar-free mentholyptus drops (2 L at 7-9 pm on the day prior to the colonoscopy with Halls®, and 2 L on the day of the colonoscopy to be completed at least 1.5 hours before the procedure with Halls®).

   ● Second arm: 2 Liters of reduced volume ascorbic acid-supplemented PEG-electrolyte (MoviPrep®) + 1 Liter of clear fluids of the patients' choice split into 2 days (1 L of MoviPrep® on the evening of the day prior to the colonoscopy + 500 mL of clear fluids of the patients choice, and another 1 L of MoviPrep® + 500 mL of clear fluids on the day of the colonoscopy to be completed at least 1 hour before the procedure.)
4. Instructions to patients:

   Patients in both arms will be instructed on how they should take the colonoscopy preparation solution, emphasizing the importance of complete intake of the solution in order to ensure a safe and effective procedure. In case of noncompliance, the remainder of the PEG solution shall be brought in by the patient for assessment. They will also be instructed to have a regular breakfast and lunch meals on the day prior to the colonoscopy, a full fluid dinner, and to stay NPO except for the colon prep after midnight till the time of colonoscopy.
5. Assessment of tolerability:

Immediately prior to the colonoscopy, patients from both study arms will be interviewed by the research coordinator to evaluate tolerability of the preparation.

Patients will be assessed for:

* Primary outcome:
* Quality of preparation: score from 1 to 4

  1. 2 3 4 Poor Fair Good Excellent
* Secondary outcome:
* Estimated volume remaining of the original PEG solution
* Palatability: score 1 to 5

  1. 2 3 4 5 Disgusting Moderately poor taste Slightly poor taste Acceptable Tasty

In addition to the following adverse events:

* Nausea
* Vomiting
* Bloating
* Cramps
* Headache
* General acceptance of the solution
* Willingness to take the preparation again in the future if necessary

VII- Sample size calculation and data analysis:

Sample size calculation was conducted based on our previously conducted study that showed a 90% good/excellent prep with Fortrans® + Halls® and the reported results on colonoscopy preparations using the reduced volume ascorbic acid-supplemented PEG-electrolyte (MoviPrep®) that range between 65-85% good/excellent (average: 75%) (1)(7-10). Therefore, based on these results and using an α of 0.05 and a power of 0.80, the sample size required to show significance was calculated to be 97 patients per arm. Hence, it was decided to recruit 100 patients per arm taking into account possible withdrawals.

For the statistical analysis, SPSS version 20.0 will be used for data entry and analysis.

The primary end point is the quality of preparation assessed by the endoscopist (who will be blind to the preparation technique). Secondary end points will be: palatability, residual volume, patient assessment of the quality of preparation, willingness to retake the preparation solution again if needed.

VIII- Study Interval:

1 year starting from the enrollment of the first patient

ELIGIBILITY:
Inclusion Criteria:

* Elective colonoscopy
* Consent to the study

Exclusion Criteria:

* Pregnant or lactating women
* Age less than 18 years
* Significant gastroparesis
* Gastric outlet obstruction
* Ileus
* Known or suspected bowel obstruction or perforation
* Phenylketonuria
* Glucose-6-phosphate dehydrogenase deficiency
* Severe chronic renal failure (creatinine clearance <30 mL/minute)
* Severe congestive heart failure (New York Heart Association [NYHA] class III or IV)
* Dehydration
* Severe acute inflammatory disease
* Compromised swallowing reflex or mental status
* Uncontrolled hypertension (SBP ≥170 mm Hg, DBP ≥100 mm Hg)
* Toxic colitis or megacolon
* Patients with IBD
* Status post partial colon resection
* Severe constipation and laxative dependent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Bowel preparation quality | 6 months
  Superiority of Fortrans + Halls to MoviPrep in cleansing the bowels

CONTACTS AND LOCATIONS:
Overall Officials: Ala I Sharara, Prof, Principal Investigator — American University of Beirut Medical Center; Fayez S Sarkis, MD, Study Director — American University of Beirut Medical Center
Locations (1):
- American University of Beirut Medical Center, Beirut, Beyrouth, Lebanon

REFERENCES:
- [Derived] Sharara AI, Harb AH, Sarkis FS, Chalhoub JM, Badreddine R, Mourad FH, Othman M, Masri O. Split-dose menthol-enhanced PEG vs PEG-ascorbic acid for colonoscopy preparation. World J Gastroenterol. 2015 Feb 14;21(6):1938-44. doi: 10.3748/wjg.v21.i6.1938. PMID 25684963